CLINICAL TRIAL: NCT02096588
Title: Detection and Prevention of Anthracycline-Related Cardiac Toxicity With Concurrent Simvastatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Principal Investigator left Johns Hopkins
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J13160; J13160 (Other: SKCCC at Johns Hopkins); NA_00091900 (Other: JHM IRB)
Record Dates: First submitted 2014-03-14; First posted 2014-03-26 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Breast cancer; Adriamycin; Simvastatin; Statin; Echocardiogram
MeSH Terms: conditions — Breast Neoplasms | interventions — Simvastatin; AC protocol; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin will be administered on an outpatient basis orally at a dose of 40 mg once daily. Treatment will start 7 days prior to the planned doxorubicin/cyclophosphamide chemotherapy initiation and will continue for a total of 25 weeks.
  Interventions: Drug: Simvastatin; Drug: Doxorubicin/cyclophosphamide
- No drug (Active Comparator): Participant not randomized to simvastatin will participate in all aspects of the study, including planned doxorubicin/cyclophosphamide chemotherapy, with the exception of simvastatin administration.
  Interventions: Drug: Doxorubicin/cyclophosphamide

INTERVENTIONS:
Drug: Simvastatin — Simvastatin will be administered on an outpatient basis orally at a dose of 40 mg once daily.
  Other Names: Zocor
  Arms: Simvastatin
Drug: Doxorubicin/cyclophosphamide — The standard chemotherapy regimen that must be planned for all participants in order to take part in this study. The regimen is given every 2 or 3 weeks per standard of care, at the direction of the treating physician.
  Other Names: Adriamycin/Cytoxan

SUMMARY:
Doxorubicin (Adriamycin), one of the drugs commonly used for the treatment of breast cancer, is in a class of medications called anthracyclines. Anthracyclines may cause heart damage that can lead to weakening of the heart muscle. This heart damage may happen right away or may occur many years after the anthracycline is given

Simvastatin is an oral medication approved by the FDA to lower cholesterol. Simvastatin is in a class of medications called statins. Some research has shown that statins may prevent heart damage that can be caused by anthracyclines like Doxorubicin (Adriamycin).

The purpose of this study is to determine if taking simvastatin while receiving the chemotherapy Doxorubicin (Adriamycin) will minimize damage to the heart.

This study is for women who will be receiving the anthracycline doxorubicin (Adriamycin) as part of their breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female Sex (Note: Patients may be pre-menopausal or post-menopausal)
* Age 18 years or older
* Histologically confirmed invasive breast carcinoma, stage I-III (Note: Estrogen Receptor (ER), Progesterone Receptor (PR) and HER2 status must be known. In newly diagnosed patients planning neoadjuvant treatment, a formal assessment of axillary lymph nodes is not required.)
* Planning to initiate adjuvant or neoadjuvant AC (adriamycin and cytoxan) chemotherapy (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 every 2-3 weeks x 4 cycles). (Note: Participants may be planning to receive adjuvant taxane therapy after the completion of AC chemotherapy. HER2 positive patients must be planning to initiate trastuzumab therapy after AC chemotherapy.)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Normal organ function and marrow function as defined by:

  * Absolute neutrophil count (ANC) ≥ 1,000
  * Platelet count ≥ 100,000
  * Total bilirubin less than or equal to the upper limit of normal
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.5 times the upper limit of normal
  * Creatinine ≤1.5 times the upper limit of normal
  * Creatine kinase (CK) ≤2.5 times the upper limit of normal
* Left ventricular ejection fraction (LVEF) as assessed by baseline echocardiogram at or above the lower limit of normal
* Women of childbearing potential must agree to use adequate contraception (non-hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of participation. Should a woman become pregnant or suspect she is pregnant while participating in the study, she should inform her treating physician immediately
* Ability to understand the study regimen and the willingness to sign a written informed consent document
* Negative pregnancy test (women of childbearing potential only)

Exclusion Criteria:

* Prior anthracycline therapy
* Currently pregnant or lactating
* Currently receiving investigational agents
* Known active liver disease (cirrhosis, chronic viral hepatitis, autoimmune liver disease or other known clinically significant active liver disease)
* Known myopathy or history of rhabdomyolysis
* Uncontrolled hypothyroidism
* History of allergic reaction or intolerance to statin treatment
* Currently receiving statin therapy or have received any statin therapy within the last 3 months
* Known history of ischemic cardiac disease (including angina requiring anti-anginal medications, myocardial infarction, coronary artery disease documented on cardiac catheterization or ischemia documented on stress test), congestive heart failure, clinically significant arrhythmia or conduction system abnormalities, clinically significant valvular disease, clinically significant pericardial effusion or EF below the lower limit of normal
* Uncontrolled inter-current illness including, but not limited to, ongoing or active serious infection, other active cardiac disease or psychiatric illness/social situations which would limit compliance with study requirements
* Inability to swallow tablets or use of a feeding tube
* Gastrointestinal disease, surgery or malabsorption that could potentially impact the absorption of the study drug
* Daily consumption of alcohol exceeding 3 standard drinks a day (defined as 10 grams of alcohol, which is equivalent to 285 mL of beer, 530 mL of light beer, 100 mL of wine or 30 mL of liquor)
* Women currently taking drugs which are strong inhibitors or inducers of CYP3A4 are not eligible. These may be found at the Indiana University Clinical Pharmacology website at http://medicine.iupui.edu/clinpharm/ddis/main-table/.
* Women taking associated with a substantial risk of myopathy when co-administered with simvastatin are not eligible. These drugs are listed in the simvastatin package insert (available at: http://www.merck.com/product/usa/pi_circulars/z/zocor/zocor_pi.pdf).
* Women taking medications for which interaction with simvastatin may result in increased levels are not eligible. Such drugs are listed in the simvastatin package insert (available at: http://www.merck.com/product/usa/pi_circulars/z/zocor/zocor_pi.pdf).
* Any medical condition which, in the opinion of the investigator, puts the patient at risk of potentially serious complications while on study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith, MD, MPH, Principal Investigator — SKCCC at Johns Hopkins
Locations (2):
- United States (2):
  - Kimmel Cancer Center at Johns Hopkins at Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 -Hopkins 7 - Sibley memorial (DC)
Pre-assignment Details: 3 subjects were screen failures, therefore 31 subjects were assigned to a treatment group in study
Period: Overall Study
Arm/Group | Simvastatin | No Drug
Started | 15 | 16
Completed | 13 | 15
Not Completed | 2 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | No Drug | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Echocardiographic Global Longitudinal Strain (GLS)
Description: To compare the absolute change in echocardiographic GLS (Global Longitudinal Strain) from baseline (T0) to 2-3 weeks after (T2) completion of 4 cycles of (neo)adjuvant anthracycline-based chemotherapy in early stage breast cancer patients who do and do not receive concurrent simvastatin therapy
Time Frame: up to 15 weeks
Population: Only participants with GLS measured on both T0 and T2 echocardiograms were evaluable for this outcome measure. Therefore, data was evaluable in only 27/31 participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change in GLS
Arm/Group | Simvastatin | No Drug
Number analyzed (Participants) | 13 | 14
Percentage change in GLS | 0.42 (2.46) | 1.11 (3.67)

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of participants with concurrent administration of simvastatin with (neo)adjuvant anthracycline-based chemotherapy in early stage breast cancer patients who experience adverse events as defined by NCI CTCAE v4.0.
Time Frame: 52 weeks
Population: Adverse event data was not collected from the "No drug" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Simvastatin | No Drug
Number analyzed (Participants) | 15 | 0
Participants | 15 |

3. Secondary Outcome: Recurrence Free Survival (RFS) With Concurrent Simvastatin
Description: To describe the recurrence free survival (RFS) in early stage breast cancer patients treated with anthracycline-based chemotherapy with and without concurrent simvastatin
Time Frame: 5 years
Population: Data was not collected
Arm/Group | Simvastatin | No Drug
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 30 days after last dose of simvastatin, up to 1 year
Description: Adverse events (AEs) were not monitored for participants in the "No Drug" arm (0 participants at risk). Only AEs possibly-related to simvastatin were recorded. The collection of toxicities related to chemotherapy and other breast cancer therapy administration was not monitored. Changes in EF or the development of other concerning findings on echocardiograms was also closely monitored.
Arm/Group | Simvastatin | No Drug
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/0
Other Adverse Events (participants affected / at risk) | 13/15 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=15) | No Drug (N=0)
CPK increased (Investigations) | 1 (1) | 0 — Elevated CK
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=15) | No Drug (N=0)
Alanine aminotransferase increased (Investigations) | 7 (10) | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Generalized Edema (General disorders) | 2 (3) | 0
Fatigue (General disorders) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT02096588/Prot_SAP_000.pdf